CLINICAL TRIAL: NCT00765349
Title: Clinical Observational Study Investigating the Role of Diastolic Dysfunction in Determining Abnormal Cardiorespiratory Exercise Testing Parameters in Patients Undergoing Major Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 08/H0902/11
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Diastolic Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients undergoing major surgery

SUMMARY:
REASON FOR STUDY

Major non-cardiac surgery has a high degree of morbidity and mortality. Recently, suitable measurements of a patient's preoperative cardiorespiratory reserve, performed non-invasively by cardiopulmonary exercise testing, have been shown to be predictive of outcome following non-cardiac surgery. Although the exact mechanisms behind poor reserve in this population are unknown, poor cardiac function and particularly diastolic dysfunction are likely to be important.

AIMS

The aim of the present study is to investigate the role of diastolic dysfunction in determining poor cardiorespiratory reserve in elderly patients undergoing major non-cardiac surgery. This will provide suitable information to inform a further therapeutic preoperative interventional study.

OBJECTIVES AND METHODS

1. To determine the presence and severity of diastolic dysfunction, measured by preoperative transthoracic echocardiogram, in a series of elderly surgical patients undergoing major elective non-cardiac surgery
2. To investigate the relationship between diastolic dysfunction and poor cardiorespiratory function during and following exercise measured by non-invasive testing including cardiopulmonary exercise testing, non-invasive blood pressure measurements and biochemical analysis
3. To determine whether patients with poor diastolic dysfunction are likely to have worse outcomes following major surgery compared with those who show no evidence of diastolic dysfunction. Outcomes will be measured in terms of length of hospital stay and early postoperative morbidity (validated scoring system) and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major surgery
* Low functional capacity

Exclusion Criteria:

* Unable to give consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing major elective surgery
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-05

CONTACTS AND LOCATIONS:
Locations (1):
- Freeman Hospital, Newcastle upon Tyne, Tyne and Wear, United Kingdom